CLINICAL TRIAL: NCT02460952
Title: The Clinic Study to Prevent Pulmonary Embolism in Patients With General Anesthesia Operation in Perioperative Period
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yingmin Ma, Vice president of Beijing Chaoyang Hospital, Beijing Chao Yang Hospital
Other Study IDs: 22704102
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism;; perioperative period;; general anesthesia
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the prevention of Pulmonary Embolism in Patients who With General Anesthesia Operation in Perioperative Period.

DETAILED DESCRIPTION:
Patients who received general anesthesia operation in Beijing Chaoyang Hospital affiliated to Capital Medical University were collected. The incidence of pulmonary embolism in perioperative period and age, gender,the surgery , clinical stage, clinical efficacy assessment will be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* The first time to accept the general anesthesia operation

Exclusion Criteria:

* Pregnancy.
* The function of liver and kidney disorder or serious abnormal electrolyte.
* The abnormal coagulation dysfunction and blood volume.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients accept Operation with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The changes of patients'Lower extremity vein in perioperative period of general anesthesia operation | 3 days before operation to 7 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: yingmin ma, doctor, Study Director — Vice president of Beijing Chaoyang Hospital
Locations (1):
- Liu Sijie, Beijing, Beijing Municipality, China